CLINICAL TRIAL: NCT03380481
Title: SouthErn China REgisTry for Stroke on Traditional Chinese Medicine
Acronym: SECRETS-TCM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yefeng Cai (Other)
Responsible Party: Sponsor-Investigator, Yefeng Cai, Director of Encephalopathy Center of Guangdong Provincial Hospital of Chinese Medcicine, Guangzhou University of Traditional Chinese Medicine
Organization: Guangzhou University of Traditional Chinese Medicine (Other)
Other Study IDs: 201604020003
Record Dates: First submitted 2017-12-13; First posted 2017-12-21 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Stroke; Cerebral Infarction; Transient Ischemic Attack; Cerebral Hemorrhage; Subarachnoid Hemorrhage
MeSH Terms: conditions — Stroke; Cerebral Infarction; Ischemic Attack, Transient; Cerebral Hemorrhage; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SECRETS-TCM: Stroke patients who treated by western medicine and/or traditional Chinese medicine in southern China
  Interventions: Other: observational only-no intervention

INTERVENTIONS:
Other: observational only-no intervention — Observational only and no predesigned interventions in this study.

SUMMARY:
Stroke is the first most common cause of death in China and one of the major causes of functional disability in the adult population.The burden of stoke is significantly increased in China in recent years.

In order to investigate the prognosis of stroke, with diagnostic and treatment information of traditional Chinese medicine (TCM), and assess the effectiveness and safety of TCM for stroke in southern China, the investigators will conduct this multicenter prospective registry study in southern China. This study will recruit 10,000 consecutive eligible patients with acute stroke from more than 50 hospitals. 24 months follow-up will be carried out on-site in hospitals and by telephone to track endpoint (including all-cause mortality, composite cerebrovascular and cardiovascular events at one and two year follow up, and neurological and functional assessments).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years.
2. Patients within 14 days of onset of acute stroke (including acute cerebral infarction, transient ischemic attack, acute cerebral hemorrhage, acute subarachnoid hemorrhage).
3. The patient and/or guardian agree to participate in this study.

Exclusion Criteria:

1. Patients with silent cerebrovascular disease.
2. Patients with non-cerebrovascular disease events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of those who meet all inclusion criteria and no exclusion criteria. Study personnel will continuously screen eligible patients presenting to the hospitals until the sample size of 10000 is reached. This study will be conducted in more than 50 hopitals in southern China.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 12 months follow-up
Composite cerebrovascular and cardiovascular events | 12 months follow-up
  Including stroke recurrence events,acute myocardial infarction and cardiac death

SECONDARY OUTCOMES:
All-cause mortality | 24 months follow-up
Composite cerebrovascular and cardiovascular events | 24 months follow-up
  Including stroke recurrence events,acute myocardial infarction and cardiac death
Modified Rankin Scale(mRS) | 3 months follow-up
  Range:Grade 0 to Grade 6, higher grade represent a worse outcome
Barthel Index(BI) | 3 months follow-up
  Range:0 to 100 points, higher points represent a better outcome
Mini-Mental State Examination(MMSE) | 3 months follow-up
  Range:0 to 30 points, higher points represent a better outcome
Modified Rankin Scale(mRS) | 12 months follow-up
  Range:Grade 0 to Grade 6, higher grade represent a worse outcome
Barthel Index(BI) | 12 months follow-up
  Range:0 to 100 points, higher points represent a better outcome
Mini-Mental State Examination(MMSE) | 12 months follow-up
  Range:0 to 30 points, higher points represent a better outcome
Modified Rankin Scale(mRS) | 24 months follow-up
  Range:Grade 0 to Grade 6, higher grade represent a worse outcome
Barthel Index(BI) | 24 months follow-up
  Range:0 to 100 points, higher points represent a better outcome
Mini-Mental State Examination(MMSE) | 24 months follow-up
  Range:0 to 30 points, higher points represent a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Yefeng Cai, M.D.,Ph D, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Wuyi Traditional Chinese Medicine Hospital of Jiangmen, Jiangmen, Guangdong, China